CLINICAL TRIAL: NCT01957332
Title: Towards Patient Tailored Cancer Treatment Supported by Molecular Imaging IMPACT: IMaging PAtients for Cancer Drug selecTion - Metastatic Breast Cancer
Brief Title: IMaging PAtients for Cancer Drug selecTion - Metastatic Breast Cancer
Acronym: IMPACT-MBC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); University Medical Center Nijmegen (Other)
Responsible Party: Principal Investigator, C.P. Schroder, MD, PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMPACT MBC
Record Dates: First submitted 2013-09-03; First posted 2013-10-08 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Breast Cancer
Keywords: molecular imaging; HER2-PET; 89Zr-trastuzumab; FES-PET; metastatic breast cancer; clinical utility
MeSH Terms: conditions — Breast Neoplasms | interventions — Molecular Imaging; proto-oncogene protein c-fes-fps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Molecular imaging (Experimental): All patients receive 18F-FES (~200MBq) injection followed by a FES-PET. On the same day or the day after 18F-FES injection 89Zr-trastuzumab (~37 MBq) will be injected. The HER2-PET will be performed 4 days after tracerinjection.
  Interventions: Procedure: Molecular imaging

INTERVENTIONS:
Procedure: Molecular imaging — On the day of FES-injection&scan or the day after FES-injection, 89Zr-trastuzumab (~37 MBq) will be injected. The HER2-PET will be performed 4 days after tracerinjection.
  Other Names: HER2-PET; Injection of 89Zr-trastuzumab followed by PET scan
Procedure: Molecular imaging — All patients receive 18F-FES (~200MBq) injection followed by a FES-PET.
  Other Names: FES injection; Injection of 18F-FES followed by PET scan

SUMMARY:
Current patient work-up, including conventional imaging and pathological assessment of just one single biopsy, might be insufficient to identify metastatic breast cancer patients, who possibly benefit from first-line anti-hormonal or anti-HER2 therapy. As receptor conversion of the tumor is found quite frequently and molecular heterogeneity can occur within one patient, up-to-date whole body information is necessary to determine estrogen receptor (ER) and/or human epidermal growth factor receptor 2 (HER2) receptor status and subsequently guide therapy decision. With molecular imaging via PET this information can be obtained in a non-invasive, patient friendly way. Furthermore, to improve and individualize treatment and be able to identify (new) drug targets and biomarkers, sampling of venous blood, circulating tumor cells (CTC), as well as circulating tumor DNA, microRNA (miRNA) and molecular characterization of one metastasis at the beginning and, if feasible, of an additional biopsy during therapy, is necessary.

DETAILED DESCRIPTION:
Patient selection for hormone therapy and anti-HER2 therapy is based on the presence of their respective targets, the ER and HER2, as currently assessed on tumor tissue by molecular biological techniques. In primary breast cancer, both ER and HER2 are powerful predictors for response to ER or HER2 targeting treatment, driving treatment decisions. If both receptors are absent, targeted hormone or anti-HER2 therapy will not be administered and chemotherapy is the only therapeutic option left. MBC management in oncology practice is often based on ER and HER2 status of the primary tumor. However, a biopsy of a metastasis is considered part of the standard work up for MBC, in view of the potential conversion of ER and HER2 during the course of the disease. In contrast to primary breast cancer, no prospective studies have been done to evaluate the impact of (converted) receptor status on metastases, on prognosis and prediction of response to subsequent targeted therapy. Although receptor conversion in MBC is a well known phenomenon, clinicians may refrain from having a biopsy taken, for instance when it would require a highly invasive procedure. Even if it is feasible, the biopsy will only reflect ER and HER2 status of a single lesion, and disregard the potential heterogeneity of expression of ER and HER2 status between and within metastatic lesions.

Therefore, the current standard work up of MBC is not adequate enough or too invasive in a relevant proportion of MBC patients to drive treatment decisions. As a result, these patients incorrectly receive an ineffective treatment with potentially toxic effects. Meanwhile, an effective treatment for these patients may be delayed or even denied (such as chemotherapy or anti-HER2 based therapy) because of inadequate assessment of ER and HER2 status. This shows the need of obtaining up-to-date whole body information with information of characteristics of the different metastases within a patient. Non-invasive 18F-fluoroestradiol(18F-FES)-PET and Zirconium-89(89Zr)-trastuzumab-PET scan techniques are able to visualize the ER and HER2 in metastatic lesions throughout the whole body, and may therefore - in a patient friendly way- provide comprehensive information (i.e. of the primary tumor and various metastatic lesions) on ER and HER2 status. Furthermore, optimal selection of the right treatment for the right patient may not only reduce unnecessary toxicity, but also health care costs. Although various studies have already indicated the clinical utility of 18F-FES-PET and 89Zr-trastuzumab-PET, no prospective data are yet available assessing their predictive value (14-19). Therefore, it is clear that these new techniques, and also the aspects of cost-effectiveness, need to be prospectively evaluated within the framework of established assessments (including metastases biopsies and FDG-PET), to ensure their implementation in standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patient with first presentation of MBC, regardless of ER and HER2 status of the primary tumor, who is eligible for first-line systemic therapy.
* Patient with non-rapidly progressive MBC, not requiring urgent initiation of chemotherapy, based on clinician's evaluation which may include:

  * no recent (< 2 weeks prior to screening visit) significant worsening of MBC related signs and symptoms according to patient history.
  * in case of liver metastases: no significant increase in liver function tests alanine aminotransferase aspartate transaminase (ASAT) and alanine transaminase (ALAT) in 2 weeks prior to screening visit. (Significant increase of liver function test is defined as 50% increase of absolute amount of ASAT/ALAT.)
* Patients in whom standard imaging work-up of MBC was recently (≤ 28 days) performed. Standard imaging must include: CT chest/abdomen, 18F-FDG-PET and bone scintigraphy.
* Patient with measurable or clinically evaluable (bone only) disease on recent standard work up of MBC are eligible.
* Metastatic lesion(s) of which a histological biopsy can safely be obtained according to standard clinical care procedures.
* Primary tumor blocks available for confirmatory central laboratory ER/HER2 testing in the UMCG. If available a snap frozen sample of the primary tumor will also be centralized in the University Medical Center Groningen (UMCG).
* WHO performance status 0-2.
* Patient is able to undergo PET imaging procedures.
* Age >18 years of age, willing and able to comply with the protocol as judged by the investigator.
* Signed written informed consent.

Exclusion Criteria:

* Contraindications for systemic treatment (as will be assigned based on biopsy and experimental scan results), either chemotherapy, hormonal therapy or anti-HER2 therapy, based on clinical judgment of treating medical oncologist and patient history.
* Pregnant or lactating women.
* Prior allergic reaction to immunoglobulins or immunoglobulin allergy.
* Inability to comply with study procedures.
* Rapidly progressive (visceral) disease requiring rapid initiation of chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2013-08-30 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Clinical utility | 3-5 years (End of study)
  The primary objective is to evaluate the clinical utility of experimental PET scans, in the setting of MBC at first presentation. These scans include Fluor-18-16 alpha-fluoroestradiol(18F-FES)-PET and Zirconium-89(89Zr)-trastuzumab-PET scans at baseline, and 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose(18F-FDG)-PET for early response measurement. Clinical utility in this setting might be defined as improved personalized medicine, when the PET scans show improved predictive value for therapy response in comparison or in addition to currently available clinical information including a biopsy. But also when the PET scans would have the same predictive value for therapy response compared to a biopsy, they would have clinical utility because they are less invasive and more patient friendly. The inherent focus (the primary endpoint) of this study is therefore therapy response. Therapy response will be related to the novel PET scans, both per patient and per metastasis analysis.

SECONDARY OUTCOMES:
Correlation PET scans & progression-free survival (PFS) | 3-5 years (End of study)
  To relate experimental PET scans (baseline 18F-FES-PET and 89Zr-trastuzumab-PET; 2 week 18F-FDG-PET scan) to (progression free) survival.
Correlation of DNA and RNA analyses to imaging, molecular analyses and follow-up data | 3-5 years (End of study)
  To relate DNA sequencing and RNA expression analysis of the baseline biopsy and venous blood samples (only DNA sequencing; baseline) to all other molecular, imaging (standard and experimental), and clinical follow-up data (treatment response and survival).
Correlation miRNA analysis to molecular analyses, imaging & clincal follow-up data | 3-5 years (End of study)
  To relate miRNA analysis of the baseline biopsy and a venous blood sample at baseline to all other molecular, imaging and clinical follow-up data.
Correlation of peptide profiling to all other molecular, imaging and clinical follow-up data | 3-5 years (EoS)
  To relate peptide profiling of new baseline biopsy and venous blood samples (baseline and day of standard response assessment) to all other molecular, imaging and clinical follow-up data.
Correlation of standard pathology results to all molecular, imaging and clinical follow up data. | 3-5 years (EoS)
  To assess molecular changes (including pathological examination) of primary biopsy, new baseline biopsy and (optional) biopsy taken during treatment and relate to all molecular, imaging and clinical follow up data.
To compare CTC enrichment approaches and correlation of CTC analysis to all molecular, imaging and clinical follow-up data | 3-5 years (EoS)
  To relate CTC count and ER/HER2 status of CTCs at baseline to all molecular, imaging and clinical follow-up data.
Correlation circulating tumor DNA analysis to all other molecular, imaging and clinical follow-up data | 3-5 years (EoS)
  To relate circulating tumor DNA analysis (baseline, day of early 18F-FDG-PET imaging and day of standard response assessment) to all other molecular, imaging and clinical follow-up data.
Cost-effectiveness of molecular imaging | 3-5 years (EoS)
  To assess cost-effectiveness of experimental PET scans.
QoL | 3-5 years (EoS)
  To assess impact of baseline biopsy procedure and baseline molecular imaging, as well as quality of Life (QoL) before and during therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Carolien Schröder, MD, PhD, Principal Investigator — University Medical Center Groningen; Willemien Menke, MD, PhD, Principal Investigator — VUMC; Winette vd Graaf, MD, PhD, Principal Investigator — RUMC
Locations (3):
- Netherlands (3):
  - VU University Medical Center, Amsterdam
  - University Medical Center, Groningen
  - University Medical Center St. Radboud, Nijmegen

REFERENCES:
- [Derived] Boers J, Eisses B, Zwager MC, van Geel JJL, Bensch F, de Vries EFJ, Hospers GAP, Glaudemans AWJM, Brouwers AH, den Dekker MAM, Elias SG, Kuip EJM, van Herpen CML, Jager A, van der Veldt AAM, Oprea-Lager DE, de Vries EGE, van der Vegt B, Menke-van der Houven van Oordt WC, Schroder CP; IMPACT-Metastatic Breast Consortium. Correlation between Histopathological Prognostic Tumor Characteristics and [18F]FDG Uptake in Corresponding Metastases in Newly Diagnosed Metastatic Breast Cancer. Diagnostics (Basel). 2024 Feb 14;14(4):416. doi: 10.3390/diagnostics14040416. PMID 38396455
- [Derived] van Geel JJL, Boers J, Elias SG, Glaudemans AWJM, de Vries EFJ, Hospers GAP, van Kruchten M, Kuip EJM, Jager A, Menke-van der Houven van Oordt WC, van der Vegt B, de Vries EGE, Schroder CP; IMPACT-Metastatic Breast Consortium. Clinical Validity of 16alpha-[18F]Fluoro-17beta-Estradiol Positron Emission Tomography/Computed Tomography to Assess Estrogen Receptor Status in Newly Diagnosed Metastatic Breast Cancer. J Clin Oncol. 2022 Nov 1;40(31):3642-3652. doi: 10.1200/JCO.22.00400. Epub 2022 May 18. PMID 35584346